CLINICAL TRIAL: NCT02953886
Title: The Effect of Silver Diamine Fluoride (SDF) on Bacteria Involved in Root or Cervical Carious Lesions Using HOMINGS Technology. A Clinical Study
Brief Title: The Effect of Silver Diamine Fluoride (SDF) on Bacteria Involved in Root or Cervical Carious Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heba Mitwalli (Other)
Collaborators: The Forsyth Institute (Other)
Responsible Party: Sponsor-Investigator, Heba Mitwalli, DDS, Master's Student, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00117560
Record Dates: First submitted 2016-10-27; First posted 2016-11-03 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Caries
Keywords: Caries; Cavity; Silver Diamine Fluoride (SDF); HOMINGS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Silver Diamine Fluoride (SDF) (Experimental): Application of Silver Diamine Fluoride (SDF) to root or cervical carious lesions (cavities). Collection of plaque pre- and one month post-SDF application.
  Interventions: Device: Silver Diamine Fluoride (SDF)

INTERVENTIONS:
Device: Silver Diamine Fluoride (SDF) — No caries removal will take place. Bacterial samples will be collected using Gracey curettes at the initial visit before application of SDF and one month after. The tooth will be dried and SDF will be placed on the carious dentin until saturated. Excess will be blotted dry with a cotton pellet
  Other Names: Silver Dental Arrest

SUMMARY:
The study will compare bacteria levels in cavities before and after silver diamine fluoride (SDF) treatment.

DETAILED DESCRIPTION:
To assess the effect of silver diamine fluoride (SDF) treatment on microorganisms present in root caries or cervical lesions by collecting microbial deposits before and 1 month after SDF application. Bacterial samples will be collected from 20 adult subjects at the initial visit before application of SDF and one month after. At the 1 month recall, examination for caries arrest will be performed. All 40 bacterial samples will be sent to the Forsyth Institute to verify bacterial composition using HOMINGS technology.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adult participants 18 years of age and older.
* At least one tooth with active (soft) cavitated lesions of ICDAS score 5 or 6 near the gingival margin (coronal cervical caries at the CEJ or exposed root surfaces with soft active carious lesions exposing dentin).

Exclusion Criteria:

* Adult participants who suffer from serious life-threatening medical diseases that interfere with basic daily self care activities.
* Patients taking antibiotics within the last two weeks.
* Patients using chlorhexidine or fluoride mouth washes within the last two weeks.
* Pregnant or breastfeeding women.
* Teeth with arrested (hard) cervical or root caries lesions.
* Teeth that have been diagnosed with an abscess or an irreversible pulpitis, or are mobile.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11; Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heba Mitwalli, DDS, Principal Investigator — University of Michigan; Margherita Fontana, DDS, PhD, Study Chair — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silver Diamine Fluoride (SDF)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Silver Diamine Fluoride (SDF)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Bacterial Composition Before and One Month After SDF Application to Root or Cervical Caries Lesions
Description: Using human oral microbiome identification using next-generation sequencing (HOMINGS), change in the total bacterial composition of all subjects was measured by the difference of the number of bacteria count from baseline to one month after SDF application.
Time Frame: baseline, One month after SDF
Measure: Number; unit: bacterial count
Arm/Group | Silver Diamine Fluoride (SDF)
Number analyzed (Participants) | 20
bacterial count
  Baseline | 1890087
  One month after SDF | 1959306

2. Primary Outcome: Caries Arrest of Teeth Measured by Change in Dentin Texture (Soft, Hard)
Description: Caries were examined for hardness or softness before and after SDF application. The change in the texture was examined after one month of SDF application the change from soft to hard is noted below.
Time Frame: One month
Measure: Number; unit: cervical lesions
Arm/Group | Silver Diamine Fluoride (SDF)
Number analyzed (Participants) | 20
cervical lesions
  Soft | 8
  Hard | 12

3. Secondary Outcome: Patient Assessment of Appearance of Treated Tooth (Concern With the Appearance of Study Tooth, Desire for the Study Tooth to be Filled)
Description: Each subject was asked if they were concerned with the appearance of the tooth that SDF was applied too. They were also asked if they wanted the study tooth to be filled with a tooth color filling.
Time Frame: One month
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride (SDF)
Number analyzed (Participants) | 20
Participants
  Concerned with appearance of tooth | 1
  Desire for tooth to be filled | 18

ADVERSE EVENTS:
Time Frame: 7 months
Description: Number of Participants at Risk is equal to the number of participants enrolled
Arm/Group | Silver Diamine Fluoride (SDF)
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silver Diamine Fluoride (SDF) (N=21)
Unfavorable taste (General disorders) | 3 (3) — When applying the SDF
Burning sensation (General disorders) | 1 (1) — When applying the SDF
Black stain (General disorders) | 21 (21) — Subjects had black stain in the cavity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT02953886/Prot_SAP_000.pdf